CLINICAL TRIAL: NCT05953675
Title: Ethanol Lock and Risk of Catheter Related Blood Stream Infection in Patients With Haemodialysis Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REG-184-2017
Record Dates: First submitted 2020-03-21; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis Catheter-Associated Bacteremia; Hemodialysis Complication
MeSH Terms: interventions — Sodium Chloride; Heparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Standard procedure of isotonic saline with heparin as lock-solution
  Interventions: Drug: Isotonic saline with heparin
- Intervention arm (Experimental): 3 mL of 70% ethanol as lock-solution
  Interventions: Drug: Ethanol 70%

INTERVENTIONS:
Drug: Ethanol 70% — Once a week, the catheter will be closed with 3 mL ethanol 70% lock-solution after a completed hemodialysis. The fluid will stay in the catheter until next hemodialysis (ca. 48 hours). The fluid will be aspirated before the hemodialysis. Standard lock-solution of isotonic saline with heparin will be used for the remaining two hemodialysis procedures of the week.
  Arms: Intervention arm
Drug: Isotonic saline with heparin — Standard procedure of isotonic saline used as lock-fluid after completed hemodialysis.
  Arms: Control arm

SUMMARY:
The aim of this study is to examine the effect of ethanol (70%) as lock-solution after hemodialysis on:

* The frequency of dialysis catheter-related bacteremia among patients under observation of potential complications
* Other complications of the use of hemodialysis-catheters eg. dysfunction of the catheter due to thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Age at or above 18 years.
* Currently recieving hemodialysis treatment with tunneled intravenous hemodialysis-catheter
* Written informed consent after verbal and written information is given.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Intolerance to ethanol or contraindications for the use of ethanol. Eg. possible interactions, former alcohol dependency.
* Earlier infections to current catheter (exit-site, tunnel-infection and catheter-related bloodstream infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Time to hemodialysis catheter-related bacteremia | 2 years

SECONDARY OUTCOMES:
Incidence of hemodialysis catheter-related bacteremia | 2 years
  number per year
Time to exit-site infection | 2 years
  days
Time to removal of catheter due to infection | 2 years
  days
Complications eg. catheter-thrombosis and pulmonary embolus | 2 years
  number per year
Life quality | 2 years
  score of QOL questionaire
Economical costs | 2 years
  Cost af treatment and cost of complications per patient year compared

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Wiese, MD,PhD, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No